CLINICAL TRIAL: NCT02392208
Title: Effect of Dialysis on the Pharmacokinetics of Telavancin in Patients With Chronic Kidney Disease Stage 5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Principal Investigator, Bruce A. Mueller, Professor and Associate Dean of Academic Affairs, College of Pharmacy, University of Michigan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00095470
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: End-Stage Renal Disease; Stage 5 Chronic Kidney Disease
Keywords: telavancin; end-stage renal disease; ESRD; pharmacokinetics; hemodialysis; chronic kidney disease; CKD; dialysis; Vibativ
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telavancin Before Hemodialysis (Other): Stage 5 Chronic Kidney Disease patients receive a single dose of telavancin before their normally scheduled hemodialysis session.
  Interventions: Drug: Telavancin; Procedure: Pharmacokinetic Blood Sampling
- Telavancin After Hemodialysis (Other): Stage 5 Chronic Kidney Disease patients receive a single dose of telavancin immediately after their normally scheduled hemodialysis session.
  Interventions: Drug: Telavancin; Procedure: Pharmacokinetic Blood Sampling

INTERVENTIONS:
Drug: Telavancin — A single 5 mg/kg dose of telavancin is administered intravenously (IV).
  Other Names: Vibativ
Procedure: Pharmacokinetic Blood Sampling — Blood samples are collected to assess telavancin plasma concentrations.
  Other Names: PK Sampling

SUMMARY:
Chronic Kidney Disease Stage 5 (CKD5) patients receiving maintenance hemodialysis are at an increased risk for developing bloodstream infections. Vancomycin is traditionally used as first-line therapy for treating these infections, but the emergence of less-susceptible bacterial strains necessitates the consideration of alternative antibiotic therapy. Telavancin is a new antibiotic that has broad-spectrum antimicrobial activity against gram-positive bacteria, including vancomycin-intermediate staphylococcus aureus. While dosing recommendations for telavancin are available for patients with normal kidney function, there are no published recommendations for CKD5 patients receiving hemodialysis. A pharmacokinetic study is needed to characterize the pharmacokinetic parameters of telavancin in these patients to determine the extent of drug removal by hemodialysis and to establish dosing recommendations for CKD5 patients on maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Within 50 - 150 % of ideal body weight and greater than 40 kg
* CKD5 receiving maintenance hemodialysis for ≥ 3 months
* Creatinine Clearance estimate < 10 mL/min
* Not received telavancin within the past month
* No concurrent illness or evidence of infection
* Able to give informed consent

Exclusion Criteria:

* Pre-study Hemoglobin < 9.0 g/dL
* Plasma Albumin < 2.5 g/dL
* Pregnancy
* Breastfeeding
* QTc interval > 470 msec on EKG obtained within the last 6 months
* Receiving concomitant QT prolonging agents
* Receiving warfarin or low molecular weight heparin products
* Known allergy to telavancin or vancomycin
* Unstable blood pressure control
* Need for routine large fluid removal during dialysis (> 4 liters)
* Diagnosis of liver disease with a Child Pugh score of C or higher
* Dialysis isolation requirements due to Hepatitis B
* Participating concurrently in another investigational drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Mueller, PharmD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Gharibian KN, Lewis SJ, Heung M, Segal JH, Salama NN, Mueller BA. Telavancin pharmacokinetics in patients with chronic kidney disease receiving haemodialysis. J Antimicrob Chemother. 2021 Dec 24;77(1):174-180. doi: 10.1093/jac/dkab370. PMID 34613416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment commenced on 07/07/15 at the University of Michigan outpatient dialysis clinics. The final participant enrolled in the study on 02/09/16.
Pre-assignment Details: All 8 participants followed a crossover study design and completed study arm 1 (telavancin before hemodialysis) followed by a 14-day minimum wash out then study arm 2 (telavancin after hemodialysis).
Groups:
- All Study Participants: Period 1: Telavancin Before Hemodialysis Stage 5 Chronic Kidney Disease patients receive a single dose of telavancin (5 mg/kg) administered intravenously (IV) before their normally scheduled hemodialysis session. Blood samples are collected over a 48-hour period to assess telavancin plasma concentrations.
  Period 2: Telavancin After Hemodialysis After a minimum 14-day period, participants from Period 1 receive another dose of telavancin (5 mg/kg). This dose is administered intravenously (IV) after the participant's normally scheduled hemodialysis session. Blood samples are collected over a 48-hour period to assess telavancin plasma concentrations.
Period: Telavancin Before Hemodialysis
Arm/Group | All Study Participants
Started | 8
Completed | 8
Not Completed | 0
Period: Telavancin After Hemodialysis
Arm/Group | All Study Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Telavancin
Description: Peak concentration of telavancin
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
mcg/mL
  Period 1: Telavancin Before Hemodialysis | 33.1 (6.8)
  Period 2: Telavancin After Hemodialysis | 38.1 (10.1)

2. Primary Outcome: Vss of Telavancin
Description: Volume of distribution of telavancin at steady state
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
mL/kg
  Period 1: Telavancin Before Hemodialysis | 201 (48)
  Period 2: Telavancin After Hemodialysis | 172 (36)

3. Primary Outcome: CLobs of Telavancin
Description: Observed clearance of telavancin
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
mL/h/kg
  Period 1: Telavancin Before Hemodialysis | 11.8 (4.6)
  Period 2: Telavancin After Hemodialysis | 6.1 (1.8)

4. Primary Outcome: t1/2 of Telavancin
Description: Half-life of telavancin
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
hours
  Period 1: Telavancin Before Hemodialysis | 13.4 (2.9)
  Period 2: Telavancin After Hemodialysis | 21.4 (5.5)

5. Secondary Outcome: AUC0-24 of Telavancin
Description: Area under the telavancin concentration-time curve 0-24 hours from start of infusion
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
mcg*h/mL
  Period 1: Telavancin Before Hemodialysis | 307 (77.1)
  Period 2: Telavancin After Hemodialysis | 465 (89.5)

6. Secondary Outcome: AUC24-48 of Telavancin
Description: Area under the telavancin concentration-time curve 24-48 hours from start of infusion
Time Frame: At hours post dose: 0, 1, 1.5, 3, 6.5, 8, 24, 48
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
mcg*h/mL
  Period 1: Telavancin Before Hemodialysis | 121 (38.3)
  Period 2: Telavancin After Hemodialysis | 220 (53.6)

ADVERSE EVENTS:
Arm/Group | Telavancin Before Hemodialysis | Telavancin After Hemodialysis
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin Before Hemodialysis (N=8) | Telavancin After Hemodialysis (N=8)
New onset atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No